CLINICAL TRIAL: NCT06136026
Title: Integrative Chinese and Western Medicine for Colorectal Cancer: A Nationwide Prospective Cohort Study
Brief Title: Integrated Chinese and Western Medicine Specialized Disease Cohort for Colorectal Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Jiangsu Famous Medical Technology Co., Ltd. (Industry)
Collaborators: Jiangsu Province Hospital of Traditional Chinese Medicine (Other); Peking University Cancer Hospital & Institute (Other); Fujian Cancer Hospital (Other Government); Hubei Cancer Hospital (Other); Shandong Cancer Hospital and Institute (Other); Shanxi Province Cancer Hospital (Other); Sichuan Cancer Hospital and Research Institute (Other); Yunnan Cancer Hospital (Other); Zhejiang Cancer Hospital (Other); Xiangya Hospital of Central South University (Other); Chongqing University Cancer Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other); First Affiliated Hospital of Guangxi Medical University (Other); First Affiliated Hospital of Harbin Medical University (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Gansu Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZLXTCXZX-2023001
Record Dates: First submitted 2023-11-06; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Cancer; Colorectal Adenoma
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, tongue coating, saliva, stool samples and tumor tissue were collected.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Rectal cancer cohort: 20,000 patients with rectal cancer will be included in this cohort and followed for five years.
- Colon cancer cohort: 20,000 patients with colon cancer will be included in this cohort and followed for five years.
- Colorectal adenoma cohort: 10,000 patients with colorectal adenomas will be enrolled in this cohort and followed for five years.

SUMMARY:
This is a nationwide cohort study on integrated traditional Chinese and Western medicine for colorectal cancer. The aim is to elucidate the distribution patterns of TCM syndromes in colorectal cancer and colorectal adenoma, reveal the relationship between TCM syndromes and diagnosis, prognosis, and prognosis. Based on biological samples, a phenotypic omics study of TCM syndromes in colorectal cancer and colorectal adenoma is conducted.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is a common malignant tumor. The global cancer data in 2020 shows that the incidence rate of CRC ranks the third in the world, and the mortality rate ranks the second in the world. China is a large country of CRC. In 2016, China's incidence rate of CRC ranked second in malignant tumors, and its mortality ranked fourth. Both incidence rate and mortality are on the rise. At present, studies have shown that TCM plays an important role in the prevention and treatment of precancerous lesions, recurrence, and metastasis of CRC throughout the entire process. However, the clinical efficacy and mechanism of TCM intervention in the onset, progression, and metastasis of CRC still need further research evidence to support. This project aims to address the above issues, based on the advantages of TCM in tumor prevention and treatment, and actively construct the first large-scale integrated traditional Chinese and Western medicine CRC specialized disease queue in China. The study focuses on the key links of the "precancerous lesions, recurrence, and metastasis" progress of CRC and conducts a combination of disease and syndrome queue research. The project is based on the team's preliminary research results and collaborates with multiple regional diagnosis and treatment centers in China to form high-quality evidence-based medical evidence and unify TCM syndrome differentiation standards for CRC. At the same time, based on the study of specialized disease cohorts, the project breaks through the phenotype omics of TCM, further revealing the biological connotation of TCM syndromes in colorectal cancer, achieving the integration of Chinese and Western medicine, breaking through the bottleneck of basic research on CRC in TCM, assisting the research process of traditional Chinese medicine in preventing and treating CRC, and promoting the modernization of TCM.

ELIGIBILITY:
Inclusion Criteria:

CRC patients:

1. The patient is over 18 years old;
2. The patient meets the diagnostic criteria for colorectal cancer;
3. The patient has not received anti-tumor treatment such as surgery, chemotherapy, radiotherapy, targeted therapy, or immunity in the past;
4. The patient voluntarily participated in this study and signed an informed consent form.

Colorectal adenoma patients

1. The patient is over 18 years old;
2. The patient meets the diagnostic criteria for colorectal adenoma;
3. The patient voluntarily participated in this study and signed an informed consent form.

Exclusion Criteria:

CRC patients:

1. Combined with other malignant tumors;
2. The patient has severe cognitive impairment, dementia, and various mental disorders.

Colorectal adenoma patients:

1. The patient had a history of malignancy;
2. The patient has severe cognitive impairment, dementia, and various mental disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnostic criteria for CRC: refer to the diagnostic criteria in the 2023 Chinese Guidelines for Integrated Diagnosis and Treatment of Malignant Tumors - Colon Cancer Part. Diagnostic criteria for colorectal adenoma: Refer to the Western diagnostic criteria for colorectal adenoma in the Pathological Diagnosis Consensus of Gastrointestinal adenoma and Benign epithelial polyps published by the Digestive Diseases Group of the Pathology Society of the Chinese Medical Association.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival of patients with CRC | 5 years
  Patients were recorded from the time they entered the study until their final death.
The detection rate of Colorectal Adenomatous Polyp. | 5 years
  In the follow-up plan, record the proportion of patients diagnosed with colorectal adenoma after colonoscopy examination.

SECONDARY OUTCOMES:
Quality of life of CRC patients | 5 years
  The quality of life will be evaluated using the KPS score. The higher the KPS score, the better the patient's health condition.
Recurrence rate of CRC patients | 5 years
  Record the number of patients with recurrence at each time point.
Metastasis rate of CRC patients | 5 years
  Record the number of patients with metastasis at each time point.
Disease-free survival (DFS) of CRC patients | 5 years
  The evaluation criteria for DFS are as follows: after radical treatment, the patient has reached a disease-free state or complete remission, and after this, the time span until the first assessment of tumor recurrence or metastasis or death without recurrence or metastasis, the patient is in a tumor free state at this stage.
Progression-free survival (PFS) of CRC patients | 5 years
  The evaluation criteria for PFS are as follows: the time span from the start of tumor treatment upon patient enrollment to the first assessment of disease progression or death without progression, during which the tumor has basically not progressed.
The canceration rate of Colorectal Adenomatous Polyp. | 5 years
  In the follow-up plan, record the proportion of patients diagnosed with colorectal cancer after colonoscopy examination.

CONTACTS AND LOCATIONS:
Overall Officials: Hai bo Cheng, Professor, Study Chair — Affiliated Hospital of Nanjing University of Chinese Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hui YF, Song SC, Zhu WJ, Bu S, Sun J, Ling TS, Cheng HB. Multicenter prospective cohort study on colorectal adenoma recurrence and malignant transformation risk based on integrative medicine: a study protocol. Front Oncol. 2025 Oct 27;15:1657390. doi: 10.3389/fonc.2025.1657390. eCollection 2025. PMID 41220937